CLINICAL TRIAL: NCT07251959
Title: Impact of Short Sessions of Exercise Therapy Plus Manual Therapy at Work on Health- and Work-related Outcomes in Office Workers With Chronic Nonspecific Spinal Pain
Brief Title: Workplace Exercise Therapy With or Without Manual Therapy in Chronic Spinal Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Murcia (Other)
Responsible Party: Principal Investigator, Martha Cecilia León Garzón, Principal Investigator, Catholic University of Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE042403
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Back Pain; Neck Pain; Low Back Pain
Keywords: Chronic nonspecific spinal pain; Exercise therapy; Sham-therapy; Massage
MeSH Terms: conditions — Back Pain; Neck Pain; Low Back Pain | interventions — Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded. Both groups will receive the same exercise sessions, delivered in small groups of up to 8 individuals that include participants from both study arms. In addition, both groups will receive a manual intervention, consisting of either manual therapy or sham manual therapy. The success of blinding will be evaluated after the intervention period by asking participants whether they believe they received the experimental intervention and how confident they are in their response (0-10 numerical rating scale).
  Because most outcomes are self-reported, effective participant blinding will also ensure blinding of outcome assessment. For muscle tone assessment, independent assessors not involved in the study will perform the measurements. Data analysts will be blinded to group allocation. Only the therapists delivering the manual therapy interventions will be aware of group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise therapy plus manual therapy (Experimental): Participants will receive 15-minute exercise therapy sessions twice per week at the workplace, including a 2-minute warm-up, 11-minute main phase, and 2-minute cool-down. The warm-up includes joint mobilization and low-load exercises. The main phase comprises six exercises in supersets, three sets of 10-12 reps with 30-second rests, divided into two blocks and targeting neck, back, and limbs, using body weight and elastic bands, with intensity rated 6-7/10 on the Borg Scale. The cool-down includes breathing and stretching exercises. Participants will also receive 15-minute manual therapy sessions twice per week, including the following myofascial techniques: nuchal ligament technique, transverse and longitudinal sliding of the paravertebral muscles on both sides of the back, and sustained pressure techniques applied to the trapezius and thoracolumbar fascia.
  Interventions: Behavioral: Exercise therapy; Procedure: Manual Therapy
- Exercise therapy plus sham manual therapy (Sham Comparator): Participants will receive the same exercise therapy protocol as the experimental group. In addition, they will receive 15-minute sham manual therapy sessions twice per week, delivered at the workplace. The sham intervention will mimic the duration, positioning, and therapist contact of the manual therapy procedures but will be applied without therapeutic intent or specific techniques to avoid producing physiological effects.
  Interventions: Behavioral: Exercise therapy; Procedure: Sham Manual Therapy

INTERVENTIONS:
Behavioral: Exercise therapy — Exercises will target the neck, upper and lower back, and upper and lower limbs, and will include military press, lateral raises, front raises, trapezius raises, rear deltoid exercise, low- and high-row exercises, good mornings with extended arms, deadlifts, squats, lunges, biceps curls, chest press, and calf raises. The protocol will be performed twice a week for 8 weeks.
Procedure: Manual Therapy — Manual therapy maneuvers twice per week for 8 weeks
  Arms: Exercise therapy plus manual therapy
Procedure: Sham Manual Therapy — Simulated manual therapy maneuvers twice per week for 8 weeks
  Arms: Exercise therapy plus sham manual therapy

SUMMARY:
Implementing workplace strategies to manage symptoms in office workers with chronic nonspecific spinal pain (CNSP) may improve both health- and work-related outcomes, as adherence to these interventions is more feasible in this context. Exercise therapy is considered the first-line treatment for CNSP; however, the added value of combining exercise therapy with manual therapy remains inconclusive. This study aims to examine the effects of short sessions of exercise therapy plus manual therapy, compared with exercise therapy plus sham manual therapy, delivered in the workplace, on health- and work-related outcomes in office workers with CNSP.

DETAILED DESCRIPTION:
Objectives: To evaluate the effects of short sessions of exercise therapy plus manual therapy compared with exercise therapy plus sham manual therapy at work on self-perceived productivity, disability, global impression of change, pain intensity, depression, anxiety, and muscle tone.

Methods: A randomized controlled trial will be conducted. The study protocol was approved by the Research Ethics Committee of Catholic University of Murcia (UCAM) (CE042403). Eligible participants will be office workers from the UCAM University with nonspecific spinal pain. Participants will be randomized into two groups. The experimental group will receive exercise therapy plus manual therapy, while the control group will receive exercise therapy plus sham manual therapy. Both groups will complete two 15-minute sessions of exercise therapy per week for 8 weeks. In addition, the experimental group will receive two 15-minute sessions of manual therapy per week, while the control group will receive sham manual therapy during the same period.

Outcomes: The primary outcomes will be self-perceived productivity, disability, patient global impression of change, and pain intensity. Secondary outcomes will include depression, anxiety, and muscle tone. Assessments will be conducted at baseline, post-intervention, and at 3- and 6-month follow-ups. Any possible adverse events will be registered during the 8-weeks of interventions.

Sample Size Estimation: Sample size was calculated using G*Power 3.1. To detect differences between groups over time, a small effect size (f = 0.17) was assumed, with 80% power and a 5% alpha level, indicating a minimum of 50 participants. Allowing for a 20% dropout rate, the target sample size was set at 60 participants (30 per group).

Statistical Analysis: A repeated-measures ANOVA (time × group) will be used. Mauchly's test will assess sphericity; if violated, the Greenhouse-Geisser correction will be applied. Post-hoc pairwise comparisons will be adjusted using Bonferroni correction. Effect sizes will be reported as partial eta-squared, and Cohen's d will be used for post-hoc comparisons. A chi-square test will assess the effectiveness of blinding by evaluating participants' perceptions of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Administrative professionals engaged in sedentary desk-based work utilizing visual display terminals (VDTs) for data processing and information management from the UCAM University
* Chronic nonspecific spinal pain defined as pain (≥4/10 on a numeric rating scale) persisting for at least the past 3 months and/or present on ≥50% of days during the previous 6 months
* The anatomical region of pain is defined from the occipital area to the gluteal folds

Exclusion Criteria:

* Participants with diagnosed conditions causing back pain, such as ankylosing spondylitis, infections, or other specific causes, including vertebral fractures
* Participants currently receiving any rehabilitative or pharmacological treatment for back pain during the 3 weeks prior to study enrollment
* Participants diagnosed with medical conditions that would prevent them from safely performing therapeutic exercise without medical supervision
* Participants who answer "Yes" to one or more questions on the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+), indicating potential contraindications to physical activity, unless cleared by a healthcare provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Work productivity and pain-related activity impairment (WPAI: Pain) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  WPAI: Pain is a self-reported instrument which assess impact of pain on work productivity and daily activities, including absenteeism, work-impairment, presenteeism, and activity-impairment
Pain intensity (Numeric Rating Scale) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  The Numeric Rating Scale (NRS) measures pain intensity on a scale from 0 (no pain) to 10 (worst possible pain), allowing self-reported assessment of pain intensity over the past week.
Patient Global Impression of Change (PGIC) | At 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  The Patient Global Impression of Change (PGIC) assesses a patient's overall perception of improvement or change in their condition since the start of treatment, using a standardized 7-point scale from 'very much improved' to 'very much worse.'
Neck Disability Index (NDI) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  Neck Disability Index (NDI) measures self-reported neck pain-related disability, including impact on daily activities, work, and function; higher scores indicate greater disability. Administered only to participants reporting neck pain
Oswestry Disability Index (ODI) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  The Oswestry Disability Index (ODI) measures self-reported disability related to low back pain, evaluating the impact on daily activities, work, and functional limitations, with higher scores indicating greater disability. Administered only to participants reporting low back pain
Adverse events | During the 8 weeks of interventions.
  Adverse events will be defined as any undesirable or harmful outcomes occurring during or after the intervention. At each exercise or manual therapy session, participants will be asked whether they have experienced any exacerbation of symptoms, including but not limited to pain, unusual fatigue, edema, tendinopathy, excessive delayed-onset muscle soreness (≥7/10), bursitis, or any other symptoms that limit or interfere with daily activities.

SECONDARY OUTCOMES:
Anxiety (GAD-7) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  The GAD-7 questionnaire assesses the severity of generalized anxiety symptoms over the past two weeks, with higher scores indicating greater anxiety levels
Severity of depressive symptoms (PHQ-9) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  The PHQ-9 questionnaire assesses the severity of depressive symptoms over the past two weeks, with higher scores indicating greater depression levels
Muscle Properties of Upper Trapezius (Myoton) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  Myoton device measures mechanical properties of skeletal muscle. Upper trapezius tone will be measured at the midpoint between the C7 spinous process and the posterior acromion border on both sides. The three firing mode will be used.
Muscle Properties of Lumbar zone (Myoton) | At baseline, 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  Myoton device measures mechanical properties of lumbar muscles. Tone will be measured 2.5 cm lateral to the L4-L5 space using the three-firing mode on both sides.

OTHER OUTCOMES:
Adequate participant blinding | At 8 weeks (end of treatment), 3 months, and 6 months post-treatment
  The success of participant blinding will be evaluated by asking participants whether they believe they received the experimental intervention and how confident they are in their response (0-10 numerical rating scale).

CONTACTS AND LOCATIONS:
Overall Officials: Martha C León-Garzón, PhD, Principal Investigator — Catholic University of Murcia
Locations (1):
- Catholic University of Murcia, Murcia, Spain